CLINICAL TRIAL: NCT00710632
Title: Predicting Weight Loss in People With Cancer: Development of a Screening Tool
Brief Title: Screening to Predict Weight Loss in Patients With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Queen's Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000590278; QMC-WEIGHT; EU-20831
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-07

CONDITIONS: Cachexia; Gastrointestinal Cancer; Hematopoietic/Lymphoid Cancer; Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: cachexia; lung cancer; gastrointestinal cancer; unspecified adult solid tumor, protocol specific; hematopoietic/lymphoid cancer
MeSH Terms: conditions — Cachexia; Gastrointestinal Neoplasms; Hematologic Neoplasms; Lung Neoplasms

INTERVENTIONS:
Other: laboratory biomarker analysis
Other: physiologic testing
Other: questionnaire administration
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Screening tests may identify people with cancer who are at high risk of losing weight and help doctors plan better treatment.

PURPOSE: This clinical trial is studying how well a new screening tool works in predicting weight loss in patients with cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify people with cancer who are at greatest risk of future weight loss by the development of a simple and practical screening tool.
* To estimate the reliability of the Appetite and Symptom Questionnaire (part 1).
* To develop a screening tool based on the ability of the optimal combination of items from the three measures (ASQ, MUST, CRP) to predict clinically significant weight loss over three months (part 2).
* To estimate the sensitivity and specificity at various cut-points of the developed screening tool in predicting clinically significant weight loss (> 10% weight loss or between 5% and 10% weight loss with a BMI < 20 kg/m^2) over three months (part 2).

OUTLINE: This is a two-part study.

* Part 1: Patients are asked to complete the Appetite and Symptom Questionnaire (ASQ) on two occasions, one week apart.
* Part 2: Patients are screened at baseline for risk of malnutrition using the Malnutrition Universal Screening Tool. Blood samples are also taken at this time to establish the level of C-reactive protein and patients complete the ASQ. Patients are weighed using calibrated scales and height measurements are obtained. Patients are asked about unplanned weight loss over the previous 3-6 months. Patients are weighed again at 3 months. Percentage weight loss is calculated at 3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria, depending on part of study:

  * Part 1:

    * Receiving radiotherapy for cancer at Nottingham City Hospital
    * Likely to be clinically stable over the duration of one week (i.e., not at high risk of disease or treatment-related appetite and weight loss)
    * Stable weight and appetite
  * Part 2:

    * Outpatient at Nottingham City Hospital with a confirmed diagnosis of primary lung or gastrointestinal cancer
    * Lost no more than 10% of pre-illness stable body weight
    * Lost no more than 5% of pre-illness stable body weight if body mass index (BMI) was less than 20 kg/m^2
    * BMI ≥ 18.5 kg/m^2

PATIENT CHARACTERISTICS:

* No condition impairing the ability to swallow
* Not receiving enteral tube feeding or parenteral nutrition (part 2)
* Able to be weighed (part 2)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent radiotherapy to the head, neck or upper gastrointestinal tract area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Percentage weight loss by measuring height and weight at baseline and at 3 months
Malnutrition Universal Screening Tool Score at initial screening
Response to the Appetite and Symptom Questionnaire at baseline
Level of blood C-reactive protein at baseline
Clinical condition, defined as diagnosis and stage of disease, treatment, and performance status at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Halliday, MSC, Principal Investigator — University of Nottingham
Locations (1):
- Queen's Medical Centre, Nottingham, England, United Kingdom